CLINICAL TRIAL: NCT04094259
Title: Proportion of the Use of Medicines and Alternative Care in Patients With Auto-Immune Diseases Alter-MAI
Brief Title: Alternative Care in Patients With Auto-Immune Diseases
Acronym: Alter-MAI
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19-0020 (ALTER-MAI)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Auto-Immune Diseases
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire. — patients will respond to a specific questionnaire regarding the use of alternative medicine

SUMMARY:
Patients followed in Internal Medicine bring together favorable conditions for the use of alternative medicines. While some are recognized for their benefits, some can, on the contrary, harm the patient. It is therefore proposed to make a complete descriptive inventory of these practices, through an anonymized questionnaire. The main objective is the evaluation of the proportion of the use of alternative medicines in patients with in the department of Internal Medicine A

DETAILED DESCRIPTION:
Patients followed in Internal Medicine department bring together favorable conditions for the use of alternative medicines. While some are recognized for their benefits, some can, on the contrary, harm the patient. It is therefore proposed to make a complete descriptive inventory of these practices, through an anonymized questionnaire. The main objective is the evaluation of the proportion of the use of alternative medicines in patients with autoimmune diseases in the department of Internal Medicine .

At all times alternative medicine has existed. Internal Medicine deals with rare autoimmune diseases, of which there is not always a cure. Even when the treatment is optimal, there are often subjective complaints.Patients followed in Internal Medicine therefore have favorable conditions for the use of alternative medicines. While some are recognized for their benefits, some can, on the contrary, harm the patient. It is therefore proposed to make a complete descriptive inventory of these practices, through an anonymized questionnaire. This information will make it possible to target the patient's needs, and to be able to offer alternative medicines that are better focused, without calling into question their conventional treatment

ELIGIBILITY:
Inclusion criteria:

* Patient with systemic lupus erythematosus (ARA and/or SLICC criteria) OR with primary Sjögren's syndrome (revised Americano European criteria) OR with systemic scleroderma (ACR/EULAR 2012 criteria)
* Patient with signed consent

Exclusion criteria:

* Patients deprived of their liberty
* Minors and adults subject to legal protection measures
* Patients subject to a justice safeguard measure
* Patient unable to understand or adhere to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with systemic lupus erythematosus (ARA and/or SLICC criteria) OR with primary Sjögren's syndrome (revised Americano European criteria) OR with systemic scleroderma (ACR/EULAR 2012 criteria)
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The number of patients using alternative medicine. | At day 1
  Counting the number of patients using alternative medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- Médecin Interne A, Limoges, France

IPD SHARING:
Plan to Share IPD: No